CLINICAL TRIAL: NCT06568679
Title: Striving for Earlier Detection and Optimization of Treatment and Prognosis for Patients With Early-onset Colorectal Cancer (EOCRC); BIO-EOCRC Study
Brief Title: Earlier Detection and Optimization of Treatment and Prognosis for Patients With Early-onset Colorectal Cancer
Acronym: BIO-EOCRC
Status: Recruiting | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: N24ECR
Record Dates: First submitted 2024-08-16; First posted 2024-08-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Early-onset Colorectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue biopsies, blood samples, stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention; observational — No intervention; observational

SUMMARY:
The study aims to collect high quality clinical data on lifestyle and patient biomaterials prior to start or during / after treatment of early-onset colorectal cancer (EOCRC) and to inform on treatment and survival outcomes of EOCRC patients.

DETAILED DESCRIPTION:
The current study will be complementary to COMPRAYA, a prospective cohort study focused on risk factors of impaired medical and psychosocial outcomes of adolescents and young adults with cancer (AYA) and to GENAYA, focused on genetic testing of AYA. The collected data and materials will be essential for an in-depth analysis of the epidemiology, exposomes and pathophysiology of EOCRC and compare this with average-onset CRC (AOCRC) and healthy controls. These data will facilitate multiomics studies and the identification of high-risk profiles and blood- and/or stool-based biomarkers, which in turn will enable the development of prevention and early detection strategies to ultimately improve prognosis and the prevalence, risk factors and mechanisms of impaired health outcomes (short- and long-term medical and psychosocial effects and late effects) over time among EOCRC patients wil be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locoregional or metastatic colorectal cancer (CRC)
* Histologically proven CRC
* Age 18 - 49 years at time of first CRC diagnosis
* Able to understand the informed consent form
* Provide written informed consent.

Exclusion Criteria:

* Mentally incompetent patients based on the opinion of treating physician
* Inability to understand the Dutch language

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with histologically proven CRC aged 18-49 years (EOCRC) are eligible for participation in this study regardless of stage and treatment of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2037-12-01 (Estimated); Study Completion 2038-12-01 (Estimated)

PRIMARY OUTCOMES:
Exploratory data analysis through a multiomics approach describing tumor biology and pathogenesis of patients with EOCRC | Change from baseline throughout follow-up of 10 years
  Associations between exposome (lifestyle factors and microbiome composition), genomics and transcriptomics and EOCRC will be determined by multivariate analysis. Multivariate tests will be applied to account for the complexity of the data and the multitude of variables involved, this will include multiple regression analysis, logistic regression analysis, and analysis of variance (ANOVA). These tests will allow us to identify and quantify the correlation between the factors and better understand the underlying mechanisms of EOCRC.

SECONDARY OUTCOMES:
Second tumor | Change from baseline throughout follow-up of 10 years
  Linkage to the Netherlands Cancer Registry (NCR) and nationwide National Pathology Database (PALGA) to asses second malignancies.
Psychological distress | Change from baseline throughout follow-up of 10 years
  Psychological distress will be assessed at each time point with the Hospital Anxiety and Depression Scale (HADS), with seven items each for assessing symptoms of anxiety and depression
Survival | Change from baseline throughout follow-up of 10 years
  Linkage will done with the Personal Records Database (BRP) to have information on survival status
Germline variants will be analysed in the carcinogenesis of EOCRC | Change from baseline throughout follow-up of 10 years
  The frequencies of germline variants that are known risk factors to cancer development will be determined. Generally, hereditary colorectal cancers will be analyzed both together with and separately from sporadic colorectal cancers. The contribution of germline variants to carcinogenesis via mutational signatures will be determined, where possible, using linear mixed models.
To compare stage-specific treatment and survival outcomes of patients with EOCRC with those of AOCRC (≥ 50 years) | Change from baseline throughout follow-up of 10 years
  Treatment and survival outcomes (progression free survival and/or recurrence free survival and overall survival) will be estimated with Kaplan-Meier curves and medians with 95% confidence intervals (CIs) will be presented and will be compared to survival outcomes of AOCRC (≥ 50 years) of a matched control group from the NCR.
High risk profiles | Change from baseline throughout follow-up of 10 years
  By a multiomics approach associations between exposomes (lifestyle, microbiome), (epi-)genomics and transcriptomics in EOCRC development and tumor phenotype will be analysed to assign high risk profiles to provide rationale for the selection of target populations that should be offered CRC screening at an earlier age.
Geno-phenotype associations | Change from baseline throughout follow-up of 10 years
  Geno-phenotype associations of patients will be analysed in-depth based on whole genome sequencing (WGS), histopathological features and survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Bolhuis, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No